CLINICAL TRIAL: NCT01470196
Title: Carfilzomib, Rituximab, and Dexamethasone (CaRD) in Waldenstrom's Macroglobulinemia
Brief Title: Carfilzomib, Rituximab and Dexamethasone in Waldenstrom's Macroglobulinemia
Acronym: CaRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-279
Record Dates: First submitted 2011-09-22; First posted 2011-11-11 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: WM; untreated; symptomatic
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Dexamethasone; Calcium Dobesilate; carfilzomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Carfilzomib, dexamethasone, rituximab
  Interventions: Drug: Dexamethasone; Drug: Carfilzomib; Drug: Rituximab

INTERVENTIONS:
Drug: Dexamethasone — 20 mg IV on Days 1, 2, 8, 9, of 21 day cycle for cycles 1-6 20 mg IV on Days 1, 2 of 21 day cycles q 2 months for cycles 1-8
  Other Names: Decadron
Drug: Carfilzomib — 20 mg/m2 IV on Days 1, 2, 8, 9 of 21 day cycles for Cycle 1 36 mg/m2 IV on Days 1, 2, 8, 9 of 21 day cycles for Cycles 2-6 36 mg/m2 IV on Days 1, 2 of 21 day cycles q 2 months for Cycles 1-8
  Other Names: PR-171
Drug: Rituximab — 375 mg/m2 IV on Days 2, 9 of 21 day cycles for Cycles 1-6 375 mg/m2 IV on Day 2 of 21 day cycles q 2 months for Cycles 1-8
  Other Names: Rituxan

SUMMARY:
Carfilzomib is a drug that has shown anti-tumor activity by inhibiting the proteasome within the cell, which is responsible for degrading or breaking down a wide variety of proteins. Carfilzomib has not been approved by the FDA.

Rituximab and dexamethasone are often used to treat Waldenstrom's Macroglobulinemia (WM), alone or in combination with other drugs. Combinations with rituximab, dexamethasone and proteasome inhibitors, like carfilzomib, show high levels of activity in WM patients.

In this research study, the investigators are testing the safety and efficacy of Carfilzomib when used along with Rituximab and Dexamethasone as a possible treatment for Waldenstrom's Macroglobulinemia.

DETAILED DESCRIPTION:
If you take part in this research study, you will receive Carfilzomib and dexamethasone as an infusion on Days 1, 2, 8, and 9 for Cycles 1-6. You will then have a Rituximab infusion on Days 2 and 9. Each cycles lasts 21 days. After completing Cycle 6 and if you are eligible, there will be a 2 month break before the maintenance phase is started. During this break, you will have a study visit with a physical exam, blood tests, and a bone marrow biopsy. If you continue to the maintenance phase, you will receive Carfilzomib and Dexamethasone on Days 1 and 2 and Rituximab on Day 2 of Cycles 1-8. Each cycle will continue to last 21 days, but will take place every 2 months. Infusions will last between 2-6 hours.

During all cycles you will have a physical exam and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. Blood tests will also be done at each Cycle visit, and you will complete a questionnaire. Bone marrow and CT scan will only be repeated at physician discretion when appropriate and in order to ensure your response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Waldenstrom's Macroglobulinemia
* Symptomatic disease
* Measurable disease
* Life expectancy of greater than 12 weeks
* Adequate organ and marrow function
* CD20 positive based on any previous performed bone marrow immunohistochemistry or flow cytometric analysis
* Disease free of prior malignancies for >/= 5 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast

Exclusion Criteria:

* More than one prior therapy
* Previous therapy with a proteasome inhibitor or rituximab
* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Currently receiving treatment for any malignancy
* Major surgery within 21 days prior to study entry
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to study entry
* Uncontrolled hypertension or uncontrolled diabetes
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to study entry
* Known history of allergy to Captisol
* Receiving any other study agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carfilzomib, rituximab, and/or dexamethasone
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating
* HIV-positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Treon, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Treon SP, Tripsas CK, Meid K, Kanan S, Sheehy P, Chuma S, Xu L, Cao Y, Yang G, Liu X, Patterson CJ, Warren D, Hunter ZR, Turnbull B, Ghobrial IM, Castillo JJ. Carfilzomib, rituximab, and dexamethasone (CaRD) treatment offers a neuropathy-sparing approach for treating Waldenstrom's macroglobulinemia. Blood. 2014 Jul 24;124(4):503-10. doi: 10.1182/blood-2014-03-566273. Epub 2014 May 23. PMID 24859363

RESULTS

PARTICIPANT FLOW:
Groups:
- Carfilzomib, Dexamethasone, and Rituximab: Carfilzomib, dexamethasone, rituximab
  Dexamethasone: 20 mg IV on Days 1, 2, 8, 9, of 21 day cycle for cycles 1-6 20 mg IV on Days 1, 2 of 21 day cycles q 2 months for cycles 1-8
  Carfilzomib: 20 mg/m2 IV on Days 1, 2, 8, 9 of 21 day cycles for Cycle 1 36 mg/m2 IV on Days 1, 2, 8, 9 of 21 day cycles for Cycles 2-6 36 mg/m2 IV on Days 1, 2 of 21 day cycles q 2 months for Cycles 1-8
  Rituximab: 375 mg/m2 IV on Days 2, 9 of 21 day cycles for Cycles 1-6 375 mg/m2 IV on Day 2 of 21 day cycles q 2 months for Cycles 1-8
Period: Overall Study
Arm/Group | Carfilzomib, Dexamethasone, and Rituximab
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate= Minor response (>25%-50% reduction in serum IgM from baseline + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Participants | 25

2. Primary Outcome: Neuropathy Incidence Rate
Description: Number and percentage of participants who experienced neuropathy attributable to CaRD therapy
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Participants | 6

3. Primary Outcome: Time to Progression
Description: Progression-free survival is the defined as the time from study entry to disease progression (PD) or death. Patients without PD are censored at the date of last disease evaluation. PD is defined as a greater than 25% increase in serum IgM and 500mg/dL absolute increase from the lowest attained response value as determined by serum electrophoresis, confirmed by at least one other investigation, or progression of clinically significant disease related symptom(s).
Time Frame: 4 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
months | 58 [9 to 65]

4. Primary Outcome: Major Response Rate
Description: Major Response Rate= Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Participants | 22

5. Primary Outcome: Very Good Partial Response and Complete Response Rate
Description: This is the rate of VGPR and CR in patients on CaRD therapy. Very good partial responses are >90% reduction in serum IgM from baseline. Complete response is defined as having resolution of all symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at every cycle visit (every 3 weeks during induction, and every 2 months during maintenance) and up to 30 days post end of treatment, up to 3 years.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=31)
Atypical chest pain (Cardiac disorders) | 1 (1) — Grade 2 unrelated atypical chest pain without evidence of arrhythmia, negative x-ray, normal troponin levels.
Pneumonia (Infections and infestations) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Grade 4 Neutrophil count decreased (Investigations) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) — Thoracic procedure complication requiring intubation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=31)
Lipase increased (Investigations) | 17
Serum amylase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 31
Peripheral Sensory Neuropathy (Nervous system disorders) | 6
Infusion related reaction (General disorders) | 8
Neutrophil count decreased (Investigations) | 11
Skin infection (Infections and infestations) | 9
Oral mucositis (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
GI cramping (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Creatinine increased (Investigations) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Platelet count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No